CLINICAL TRIAL: NCT04892576
Title: Stretch-shortening Cycle Exercises: an Efficient Training Model for Optimizing Gait-symmetry and Balance Capabilities in Children With Unilateral Cerebral Palsy
Brief Title: Strength Training in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0018/0078
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: A prospective pre-test post-test randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participants in this group received the standard physical rehabilitation program.
  Interventions: Other: Physical Therapy
- SSC group (Experimental): Participants in this group received the standard physical rehabilitation program as the control group in addition to the SSC exercise program
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — The control group recieved the standard physical rehabilitation program conducted for 45 minutes, twice a week for eight consecutive weeks, and consisted of advanced balance training, gait training, postural and flexibility exercises, and strength training exercises.
  The SSC group received the same program in addition to the SSC exercises for 30 minutes, two times per week for eight successive weeks

SUMMARY:
This study was set out to assess the effect of stretch-shortening (SSC) exercises on gait-symmetry and balance in children with unilateral cerebral palsy (UCP). Forty-two children with UCP were randomly allocated to the control group (n = 21, received standard physical rehabilitation) or the SSC group (n =21, received standard rehabilitation plus SSC exercises). Both groups were assessed for ait-symmetry and balance pre and post-treatment.

DETAILED DESCRIPTION:
Forty-two children with UCP were recruited from the Physical Therapy Outpatient Clinic of Collee of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, King Khalid Hospital, and a tertiary referral hospital, Al-Kharj, Saudi Arabia. Their age ranged between 8 and 12 years, were functioning at levels I or II according to the Gross Motor Function Classification System, and had spasticity level 1 or 1+ per the Modified Ashworth Scale. Children were excluded if they had fixed deformities, underwent neuromuscular or orthopedic surgery in the last 12 months, submitted to BOTOX injection in the past 6 months, attentional neglect, cardiopulmonary problems preventing them from performing high-intense exercise training.

Outcome measures

1. Gait-symmetry Indices: Gait symmetry indices (Spatial and temporal) were measured through a 3D motion analysis system.
2. Balance capabilities: several aspects of balance including sensory organization, reactive balance, and rhythmic weight shift were tested through a Pro Balance Master system.

The control and SSC groups received a standard rehabilitation program for 45 minutes, twice a week for eight consecutive weeks. The program comprised advanced balance training, and gait training exercises, postural and flexibility exercises, strength training exercises. Additionally, the SSC group received an SSC exercise program for 30 minutes, twice/week for eight weeks per the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The SSC program consisted of ten unilateral and bilateral lower limb plyometrics in the form of hopping/bounding/jumping activities. The SSC training was preceded by a warm-up for 5 minutes and ended up with a 5-min cooldown.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cerebral palsy
* age from 8 to 12 years
* motor function level I or II according to the Gross Motor Function Classification System
* Spasticity level 1 or 1+ according to the Modified Ashworth Scale

Exclusion Criteria:

* Structural deformities
* Musculoskeletal or neural surgery in the last year
* BOTOX injection in the last 6 months.
* cardiopulmonary disorders interfering with the ability to engage in exercise training
* hemispatial neglect

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Gait symmetry | 2 months
  Gait symmetry indices (spatial and temporal) were measured about the step length and single-limb support time of the paretic and non-paretic leg through a 3D motion analysis system
Balance Capabilities | 2 months
  Some aspects of balance capabilities including sensory organization, reactive balance, and rhythmic weight shift were measured through a Pro Balance Master sytem.

CONTACTS AND LOCATIONS:
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No